CLINICAL TRIAL: NCT02708732
Title: UK Utility Study in Diffuse Large B-Cell Lymphoma
Brief Title: Utility Study in Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29956
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- DLBCL Participants: A cohort of approximately 100 patients in first remission with DLBCL will complete questionnaires through a 15-minute postal or online survey.

SUMMARY:
This study is a prospective, cross-sectional survey to be administered to real patients in remission from DLBCL using a 15-minute postal or online survey. The project is designed to describe the impact of DLBCL remission on health utility and quality of life. Data collection will occur over a 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (>/=) 18 years of age
* Diagnosis of DLBCL and currently in first remission
* Prior drug treatment for DLBCL

Exclusion Criteria:

* Receiving active treatment for DLBCL
* Relapsed following any treatment for DLBCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 patients in first remission with DLBCL will be recruited from online advertisements and a specialist medical recruitment agency to complete study-administered questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life According to European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) Score | Up to 4 months of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PH Associates - an OPen Health Company, Marlow, United Kingdom